CLINICAL TRIAL: NCT01178554
Title: Child System and Treatment Enhancement Projects (Child STEPs); The Clinic Treatment Project - Phase II
Brief Title: The Clinic Treatment Project
Acronym: CTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Judge Baker Children's Center (Other)
Collaborators: MacArthur Foundation (Other); University of Hawaii (Other); University of Illinois at Chicago (Other)
Responsible Party: John R. Weisz, Judge Baker Children's Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 83423-0
Record Dates: First submitted 2010-07-12; First posted 2010-08-10 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Anxiety; Depression; Problem Behavior
Keywords: anxiety disorders; depression; depressive disorders; disruptive behavioral problems; conduct problems
MeSH Terms: conditions — Anxiety Disorders; Depression; Problem Behavior; Depressive Disorder | interventions — Psychotherapy; Therapeutics; Case Management; Practice Guidelines as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care Treatment (Active Comparator): Usual Care therapists could use any treatment procedures they used regularly in their clinical practice.
  Interventions: Behavioral: psychotherapy
- Standard Manual Treatment (SMT) (Experimental): Evidence-based treatment manuals were used for anxiety (Coping Cat Manual; Kendall, 1994; Kendall et al., 1994 ), depression (Primary and Secondary Control Enhancement Training; Weisz et al., 1997, 1998), and conduct problems (Defiant Children Manual; Barkley, 1997).
  Interventions: Behavioral: evidence-based treatment
- Modular Maual Treatment (MMT) (Experimental): Therapists used a modular manual (Modular Approach to Therapy for Children with Anxiety, Depression, or Conduct Problems; Chorpita & Weisz, 2004) to help children with primary problems of anxiety, depression, and conduct.
  Interventions: Behavioral: modular evidence-based treatment

INTERVENTIONS:
Behavioral: psychotherapy — Usual Care therapists could use any treatment procedures they used regularly in their clinical practice.
  Other Names: Treatment As Usual (TAU); Case Management
  Arms: Usual Care Treatment
Behavioral: evidence-based treatment — Evidence-based treatment manuals were used for anxiety (Coping Cat Manual; Kendall, 1994; Kendall et al., 1994 ), depression (Primary and Secondary Control Enhancement Training; Weisz et al., 1997, 1998), and conduct problems (Defiant Children Manual; Barkley, 1997).
  Other Names: best practices; evidence-based practices; treatment manuals
  Arms: Standard Manual Treatment (SMT)
Behavioral: modular evidence-based treatment — Therapists used the Modular Approach to Therapy for Children with Anxiety, Depression, or Conduct Problems (MATCH-ADC; Chorpita & Weisz, 2004)
  Other Names: modular treatments; best practices; evidence-based practices
  Arms: Modular Maual Treatment (MMT)

SUMMARY:
The Clinic Treatment Project tested two alternative methods of delivering evidence-based practices within public community-based mental health clinics, using training and supervision procedures designed for the settings and users.

DETAILED DESCRIPTION:
The Clinic Treatment Project focused on ethnically diverse youths aged 7-13 who were referred to community-based mental health clinics for problems involving disruptive behaviors, depression, anxiety, and any combination of these. Using a randomized block design, therapists were randomly assigned to deliver usual treatment procedures (usual care, or UC) in their clinics or evidence-based practices deployed in two forms: (a) standard manual treatment (SMT), using full treatment manuals, one at a time, exactly as they have been tested in clinical trials, and (b) modular manual treatment (MMT) in which therapists learn the component practices of the standard manuals but individualize the use of the components for each child using a guiding clinical algorithm. Unlike the SMT approach, the MMT approach allows the duration and sequencing of techniques to be individualized in an effort to fit the child's needs and allows the clinician to draw techniques from outside the target disorder domain when needed (e.g., to address noncompliance during the course of treating depression). Both SMT and MMT were supported by training and supervision procedures designed to fit providers and their clinic contexts. Assessments were carried out at pre-treatment, at post-treatment, and at 3-, 6-, 9-, 12-, 18-, and 24-month follow-ups. Assessments carried out at pre-treatment included(a) individual youth problems and disorders; (b) individual youth functioning at home and school; and (c) clinic staff beliefs and attitudes toward their work and workplace. Assessments carried out at post-treatment and follow-up only included measures of (a) youth, parent, and therapist satisfaction with treatment; (b) youth, parent and therapist views on the quality of the therapeutic relationship; and (c) treatment costs. Assessments carried out at follow-up only included (a) parent reports of any mental health service use following project treatment, and (b) therapist reports on the extent to which the treatment procedures they used in the project are continued after project termination. Analyses will address critical questions about deployment of evidence-based youth practices to clinical care settings.

ELIGIBILITY:
Inclusion Criteria:

* 7 - 13 year olds and their parents
* seeking services at community mental health clinics
* primary problem or disorder related to anxiety, depression, or conduct problems

Exclusion Criteria:

* Child is younger than 7 years, 9 months or older than 13 on the day of the phone screen.
* Child has attempted suicide within the past year.
* Schizophrenic spectrum diagnosis (including MDD w/ psychotic features)
* Autism or another Pervasive Developmental Disorder (e.g., PDD NOS, Asperger's Disorder, Child Disintegrative Disorder, Rett's Disorder).
* Anorexia Nervosa
* Bulimia Nervosa
* Mental Retardation
* No relevant T-scores validate target disorders.
* ADHD identified as primary reason for seeking treatment at phone screen
* Child's sibling already included
* Child's medication has not been regulated for one month or longer

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2005-06; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Brief Problem Checklist (BPC, parent and child forms) | Change over time from Day 1 to Day 267
  Youth and parents were contacted weekly to report changes in youth functioning. Each person was asked to rate their own or their child's behavior on 12 items (6 internalizing and 6 externalizing behaviors) that were adapted from the Youth Self Report and the Child Behavior Checklist. Children and caregivers completed the pre-treatment assessment on Day 1, every week during treatment, and at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment.

SECONDARY OUTCOMES:
The Children's Interview for Psychiatric Syndromes-Child and Parent Forms (ChIPS/P-ChIPS) | Change over time from Day 1 to Day 267
  The ChIPS/P-ChIPS are structured psychiatric interviews designed to assess psychopathology according to DSM-IV criteria in children and adolescents ages 6-18 years. ChIPS/P-ChIPS assess twenty behavioral, anxiety, mood, and other syndromes as well as psychosocial stressors the child might have experienced. Symptoms are assessed using a "yes/no" question format. Onset, offset and duration data are gathered for each disorder. On average, youth and caregivers completed the post-treatment assessment 267 days (SD=124 days) after the pre-treatment assessment.(Used as a measure of clinical outcome.)
Top Problems Assessment | Change over time from Day 1 to Day 712 (24-mo follow-up)
  Youths and parents were asked to identify "The three most important problems for which you need [or "your child needs"] help." at the intake assessment. The six resulting problems (3 from youth, 3 from parent) were then rated on a scale of 0 ("Not serious at all") to 10 ("Very serious problem") by youth and parent. Youths and parents completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1. (Used as a measure of clinical outcome.)
Youth Self-Report Form (YSR) | Change over time from Day 1 to Day 712 (24-mo follow-up)
  The YSR assesses problems in children on eight narrow-band scales (Withdrawn, Somatic Complaints, Anxious, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, Aggressive Behavior), three broad-band scales (Internalizing, Externalizing, and Total problems), and six DSM-oriented scales. Children completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1.(Used as a measure of clinical outcome.)
Child Behavior Checklist (CBCL) | Change over time from Day 1 to Day 712 (24-mo follow-up)
  The CBCL assesses problems in children on eight narrow-band scales (Withdrawn, Somatic Complaints, Anxious, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, Aggression), three broad-band scales (Internalizing, Externalizing, and Total problems), and six DSM-oriented scales. Caregivers completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1. (Used as a measure of clinical outcome.)
Therapeutic Alliance Scale for Children | post-treatment (Day 267)
  The quality of youths' working alliance with their therapists was assessed via the Therapeutic Alliance Scale for Children (TASC, Shirk & Saiz, 1992). The 7-item scale comes in both a youth-report form and a parent-report form (parents reporting on their youth's relationship with the therapist). On average, children and caregivers completed the post-treatment assessment 267 days (SD = 124 days) after the pre-treatment assessment. (Available for supplemental analyses.)
Service Assessment for Children and Adolescents: Treatment and Auxiliary Service Use Scales | Change over time from Day 1 to Day 712 (24-mo follow-up)
  The SACA (Horwitz et al., 2001)is a standardized interview for youths and parents that measures use of mental health services across a broad spectrum (including outpatient, inpatient, and school-based). SACA reliability and validity data are well-documented. Caregivers completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 12- and 24-month follow-up from Day 1.(Available for supplemental analyses.)
Revised Children's Anxiety and Depression Scale | Change over time from Day 1 to Day 267
  The RCADS is a 47-item child self-report measure that assesses symptoms of several DSM-IV anxiety and depressive disorders (i.e., separation anxiety disorder, social phobia, obsessive-compulsive disorder, panic disorder, generalized anxiety disorder, and major depressive disorder). On average, children and caregivers completed the post-treatment assessment 267 days (SD = 124 days) after the pre-treatment assessment.(Available for supplemental analyses.)
Brief Symptom Inventory | Change over time from Day 1 to Day 267
  The Brief Symptom Inventory (BSI) is a parent self-report form that is the short form of the Symptom Checklist-90 Revised instrument. The BSI provides a screen for psychological problems. This inventory reports profiles of nine primary symptom dimensions and three global indices of distress (Derogatis, 1993). It can also be used to measuring patient progress during treatment or in the assessment of treatment outcomes. On average, caregivers completed the post-treatment assessment 267 days (SD = 124 days) after the pre-treatment assessment. (Available for supplemental analyses.)
Brief Impairment Scale | Change over time from Day 1 to Day 712 (24-mo follow-up)
  The BIS is a 23-item instrument that evaluates three domains of functioning: interpersonal relations, school/work functioning, and self-care/self-fulfillment. Its advantages over other global impairment instruments are that it is respondent based, short in administration time, and multidimensional. Caregivers completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 12- and 24-month follow-up from Day 1.(Available for supplemental analyses.)
Services for Children & Adolescents - Parent Interview (SCAPI) | Change over time from Day 1 to Day 712 (24-mo follow-up)
  The SCAPI is a measure that tracks child's use of medication as reported by the parent. Caregivers completed the pre-treatment assessment on Day 1, at post-treatment assessment which occurred on average 267 days (SD = 124 days) after the pre-treatment assessment, and at 3-, 6-, 9-, 12- and 24-month follow-up from Day 1.(Available for supplemental analyses.)

CONTACTS AND LOCATIONS:
Overall Officials: John R. Weisz, Ph.D., Principal Investigator — Judge Baker Children's Center; Bruce F. Chorpita, Ph.D., Principal Investigator — University of Hawaii
Locations (2):
- United States (2):
  - The University of Hawaii at Manoa, Honolulu, Hawaii
  - Judge Baker Children's Center, Boston, Massachusetts

REFERENCES:
- [Background] Chorpita BF, Bernstein A, Daleiden EL; Research Network on Youth Mental Health. Driving with roadmaps and dashboards: using information resources to structure the decision models in service organizations. Adm Policy Ment Health. 2008 Mar;35(1-2):114-23. doi: 10.1007/s10488-007-0151-x. Epub 2007 Nov 6. PMID 17987376
- [Background] Borntrager CF, Chorpita BF, Higa-McMillan C, Weisz JR. Provider attitudes toward evidence-based practices: are the concerns with the evidence or with the manuals? Psychiatr Serv. 2009 May;60(5):677-81. doi: 10.1176/ps.2009.60.5.677. PMID 19411357
- [Background] Ebesutani C, Bernstein A, Nakamura BJ, Chorpita BF, Higa-McMillan CK, Weisz JR; The Research Network on Youth Mental Health. Concurrent Validity of the Child Behavior Checklist DSM-Oriented Scales: Correspondence with DSM Diagnoses and Comparison to Syndrome Scales. J Psychopathol Behav Assess. 2010 Sep;32(3):373-384. doi: 10.1007/s10862-009-9174-9. Epub 2009 Nov 27. PMID 20700377
- [Background] Chorpita BF, Reise S, Weisz JR, Grubbs K, Becker KD, Krull JL; Research Network on Youth Mental Health. Evaluation of the Brief Problem Checklist: child and caregiver interviews to measure clinical progress. J Consult Clin Psychol. 2010 Aug;78(4):526-36. doi: 10.1037/a0019602. PMID 20658809
- [Background] Ebesutani C, Bernstein A, Nakamura BJ, Chorpita BF, Weisz JR; Research Network on Youth Mental Health. A psychometric analysis of the revised child anxiety and depression scale--parent version in a clinical sample. J Abnorm Child Psychol. 2010 Feb;38(2):249-60. doi: 10.1007/s10802-009-9363-8. PMID 19830545
- [Background] Ho A, Weisz JR, Austin AA, Chorpita BF, Southam-Gerow M, Wells K, the Research Network on Youth Mental Health. Bridging science and community practice: Clinician and organizational engagement in community clinics in the clinic treatment project. Emotional and Behavioral Disorders in Youth. Winter 2006;7:13-19.
- [Background] Martin JL, Weisz JR, Chorpita BF, Higa CK, Southam-Gerow M, Wells K, the Research Network on Youth Mental Health. Moving evidence-based practices into everyday clinical care settings: Addressing challenges associated with pathways to treatment, child characteristics, and structure of treatment. Emotional and Behavioral Disorders in Youth. Winter 2006;7:5-21.
- [Background] Palinkas LA, Aarons GA, Chorpita BF, Hoagwood K, Landsverk J, Weisz JR; Research Network on Youth Mental Health. Cultural exchange and the implementation of evidence-based practice: two case studies. J Evidence-Based Social Work. 2009 September;19(5):602-612.
- [Background] Palinkas LA, Schoenwald SK, Hoagwood K, Landsverk J, Chorpita BF, Weisz JR; Research Network on Youth Mental Health. An ethnographic study of implementation of evidence-based treatments in child mental health: first steps. Psychiatr Serv. 2008 Jul;59(7):738-46. doi: 10.1176/ps.2008.59.7.738. PMID 18586990
- [Derived] Weisz JR, Chorpita BF, Palinkas LA, Schoenwald SK, Miranda J, Bearman SK, Daleiden EL, Ugueto AM, Ho A, Martin J, Gray J, Alleyne A, Langer DA, Southam-Gerow MA, Gibbons RD; Research Network on Youth Mental Health. Testing standard and modular designs for psychotherapy treating depression, anxiety, and conduct problems in youth: a randomized effectiveness trial. Arch Gen Psychiatry. 2012 Mar;69(3):274-82. doi: 10.1001/archgenpsychiatry.2011.147. Epub 2011 Nov 7. PMID 22065252
- See also: Child System and Treatment Enhancement Projects — http://www.child-steps.org/